CLINICAL TRIAL: NCT06150950
Title: RCT of the Effects of Cardiac reHABilitation (REHAB) Among Patients With Fontan Failure
Brief Title: REHAB Fontan Failure: A Trial of Cardiac Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Vanderbilt University Medical Center (Other); Adult Congenital Heart Association (Unknown); Julie Fletcher Memorial Fund (Unknown); Pete Huttlinger Memorial Fund (Unknown)
Responsible Party: Principal Investigator, Daniel Clark, Assistant Professor of Adult and Pediatric Cardiology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 67788
Record Dates: First submitted 2023-05-30; First posted 2023-11-30 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure Congenital; Single-ventricle
Keywords: Fontan; Single ventricle; Cardiac rehabilitation
MeSH Terms: conditions — Univentricular Heart | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Intervention Model Description: At enrollment, participants will be randomized in a 1:1 ratio to cardiac rehabilitation or usual care using randomly permuted blocks of 2, 4, and 6. The randomization will be stratified by study site and time from Fontan palliation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiac rehabilitation (Experimental): For patient randomized to cardiac rehabilitation, the ACHD clinician will place the referral after they and the patient have seen the group assignment. All participants will be referred to Heart Fit for Life community-based cardiac rehabilitation program in Palo Alto, CA. Cardiac rehabilitation will be offered as an in-person, hybrid, or completely virtual program for Stanford participants and will be entirely virtual for Vanderbilt participants. Participants will attend 3 sessions per week for 12 weeks. Participants will receive weekly email reminders via the electronic medical record to encourage participation. The study protocol pertains only to referral to cardiac rehabilitation. All other aspects of the cardiac care will be at the discretion of clinicians. All study participants will receive a Fitbit for daily activity tracking.
  Interventions: Behavioral: Cardiac rehabilitation
- Usual care (Active Comparator): For patients randomized to the usual care (no cardiac rehabilitation group), cardiac rehabilitation will not be initiated between randomization and for up to 16 weeks following randomization. The study protocol controls only referral to cardiac rehabilitation. All other aspects of the cardiac care, such as titration of guideline directed medical therapy will be at the discretion of clinicians. All study participants will receive a Fitbit for daily activity tracking.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Cardiac rehabilitation — Cardiac rehabilitation is a multifaceted, comprehensive therapeutic intervention of personalized, supervised exercise training that is beneficial and well-studied among patients with non-ACHD heart failure and has consistently been shown to improve QOL. Unfortunately, cardiac rehabilitation has been underutilized with an overall participation <50% of eligible patients despite international guidelines advocating for more consistent deployment of cardiac rehabilitation. A major a barrier to cardiac rehabilitation is access, as CMS-mandates a physician be within 3 minutes of the rehabilitation facility to assure insurance reimbursement. This mandate limits isolated, outpatient cardiac rehabilitation programs, especially in rural communities.
  Arms: Cardiac rehabilitation
Other: Usual care — For participants randomized to the usual care (no cardiac rehabilitation group), cardiac rehabilitation will not be initiated between randomization and for up to 16 weeks following randomization. The study protocol controls only referral to cardiac rehabilitation. All other aspects of the cardiac care, such as titration of guideline directed medical therapy will be at the discretion of clinicians.
  Arms: Usual care

SUMMARY:
The goal of this clinical trial is to compare the impact of cardiac rehabilitation on Fontan failure patients' exertional tolerance, frailty, and quality of life.

1. Among patients with Fontan failure, will cardiac rehabilitation increase average daily steps compared to usual care?
2. Among patients with Fontan failure, will cardiac rehabilitation improve exertional tolerance (as measured by cardiopulmonary exercise testing), frailty, and self-reported quality of life metrics compared to usual care?

DETAILED DESCRIPTION:
REHAB Fontan Failure is a a multi-center, non-blinded, randomized clinical trial evaluating the effect of cardiac rehabilitation compared to usual care on exercise tolerance among adults with Fontan failure. Eligible study subjects will be identified from clinical chart review and study informational fliers will be sent to Adult Congenital Heart Disease (ACHD) cardiologists at all centers. Fontan failure patients being evaluated for outpatient care at ACHD centers and meeting eligibility criteria will be enrolled and randomly assigned to either cardiac rehabilitation or usual clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Fontan failure, defined as history of a Fontan procedure and at least one of the following: systemic ventricular EF <50% (by echocardiography, cardiac magnetic resonance imaging, or computer tomography), protein losing enteropathy, plastic bronchitis, chronic loop diuretics prescribed by ACHD Cardiologist, and/or peak VO2 < 50% predicted (by FRIEND equation)
* Age >= 18 years old

Exclusion Criteria:

* Inotrope-dependence
* Symptomatic, uncontrolled arrhythmias
* Pregnancy
* Contraindication to cardiac rehab or already enrolled in cardiac rehabilitation
* Inability to comply with the protocol
* Recent (<3 months) planned Fontan pathway percutaneous or surgical intervention
* Resting hypoxemia with baseline oxygen saturation <80%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Average daily step count | 120 days (+/- 45 days) post-randomization
  Average daily step count during the intervention period measured by Fitbit 3 activity tracker

SECONDARY OUTCOMES:
Change in 5-meter timed walk as a measure of slowness | Baseline and 120 days (+/- 45 days) post-randomization
Change in exercise time as a measure of exhaustion | Baseline and 120 days (+/- 45 days) post-randomization
  Exercise time on cardiopulmonary exercise testing
Change in respiratory exchange ratio (RER) as a measure of exhaustion | Baseline and 120 days (+/- 45 days) post-randomization
  RER on cardiopulmonary exercise testing (exhaustion)
Change in mini-nutritional assessment short form (MNA-SF) score | Baseline and 120 days (+/- 45 days) post-randomization
  Nutrition score as measured by MNA-SF; range 0-14; malnourished 0-7, 8-11 at-risk, and 12-14 normal nutritional status
Change in body fat percentage | Baseline and 120 days (+/- 45 days) post-randomization
  Body fat percentage is a measure of body composition
Change in grip strength | Baseline and 120 days (+/- 45 days) post-randomization
Change in patient reported physical activity questionnaire score | Baseline and 120 days (+/- 45 days) post-randomization
  The physical activity questionnaire score ranges from 0 - 10,000 kilo-calories/week, with higher scores representing higher physical activity.
Change in Kansas City Cardiomyopathy Questionnaire-12 (KCCQ-12) scale score | Baseline and 120 days (+/- 45 days) post-randomization
  KCCQ-12 is a 12 question questionnaire, participants completed questionnaire about how heart failure affected their life over the past 2 weeks. The scale has 4 domains: symptom frequency, physical limitation, social limitations and quality of life for a total possible transformed score of 0 to 100 where 100 denotes the highest health status. A positive change from baseline indicates improvement.
Change Patient Health Questionnaire-2 (PHQ-2) score | Baseline and 120 days (+/- 45 days) post-randomization
  Mood assessment (Range 0-6, higher score indicates higher risk of depression, >=3 suggestive of depression)
Average daily active minutes | Baseline and 120 days (+/- 45 days) post-randomization
  Total average daily active minutes from Fitbit
Average daily active minutes of moderate-high intensity activity | Baseline and 120 days (+/- 45 days) post-randomization
  Average daily active minutes of moderate-high intensity activity from Fitbit
Average daily sedentary minutes | Baseline and 120 days (+/- 45 days) post-randomization
  Average daily sedentary minutes from Fitbit
Change in peak respiratory oxygen uptake (VO2) | Baseline and 120 days (+/- 45 days) post-randomization
  Peak VO2 on follow-up cardiopulmonary exercise testing, adjusted for baseline
Change in oxygen (O2) pulse | Baseline and 120 days (+/- 45 days) post-randomization
  O2 pulse on follow-up cardiopulmonary exercise testing, adjusted for baseline
Change in minute ventilation/carbon dioxide production (VE/VCO2) | Baseline and 120 days (+/- 45 days) post-randomization
  VE/VCO2 on follow-up cardiopulmonary exercise testing, adjusted for baseline
Change in anaerobic threshold | Baseline and 120 days (+/- 45 days) post-randomization
  Anaerobic threshold on follow-up cardiopulmonary exercise testing, adjusted for baseline

OTHER OUTCOMES:
Exploratory outcome: number of participants with exercise-induced clinical ailment | 120 days (+/- 45 days) post-randomization
  Sustained arrhythmia or hemodynamic change necessitating hospitalization, heart failure hospitalization, or all-cause death within 30 days of completion of cardiac rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E Clark, MD, MPH, Principal Investigator — Stanford University; Jonathan N Menachem, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No